CLINICAL TRIAL: NCT07392918
Title: Esophageal Pressure-guided Personalized Recruitment Pressure During Pneumoperitoneum in Trendelenburg Position Laparoscopy: A Prospective Randomized Controlled Trial
Brief Title: Esophageal Pressure-guided Personalized Recruitment Pressure During Pneumoperitoneum in Trendelenburg Position Laparoscopy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ju Gao (Other)
Responsible Party: Sponsor-Investigator, Ju Gao, Study Director, Northern Jiangsu People's Hospital
Organization: Northern Jiangsu People's Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: 2026KY021
Record Dates: First submitted 2026-01-31; First posted 2026-02-06 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Pressure; Recruitment Maneuver
Keywords: Esophageal Pressure; Recruitment Maneuver; Trendelenburg Position; Laparoscope

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Personalized Lung Recruitment Pressure Group (Experimental): The inspiratory and expiratory esophageal pressures (Pes) are measured using a transnasal esophageal balloon catheter to estimate pleural pressure, thereby calculating the transpulmonary pressure in the non-dependent lung regions. Under conditions of homogeneous lung parenchyma, the physiological upper limit of transpulmonary pressure is 20 cmH₂O. To achieve this upper limit at end-inspiration in the non-dependent lung tissue, the lung recruitment pressure(P) is calculated with the formula: P = 20 × ΔP / [ΔP - (Pes_insp - Pes_exp)], where the maximum pressure does not exceed 40 cmH₂O;ΔP is Driving Pressure. Using the calculated pressure, a single-cycle recruitment maneuver is performed both 30 minutes after pneumoperitoneum establishment and before the end of surgery, each maintained for 10 seconds.
  Interventions: Procedure: Esophageal Pressure
- Fixed Lung Recruitment Pressure Group (Other): A single-cycle lung recruitment maneuver was performed at a fixed pressure of 30 cmH₂O for 10 seconds, both 30 minutes after pneumoperitoneum establishment and immediately before the end of surgery.
  Interventions: Procedure: Lung Recruitment Maneuver

INTERVENTIONS:
Procedure: Esophageal Pressure — A transnasally placed esophageal balloon catheter was inserted. Following a positive-pressure occlusion test, end-inspiratory and end-expiratory esophageal pressures (Pes) were measured to estimate pleural pressure, thereby enabling the calculation of transpulmonary pressure in the non-dependent lung regions.Under conditions of homogeneous lung parenchyma, the physiological upper limit of transpulmonary pressure is 20 cmH₂O. To achieve this upper limit at end-inspiration in the non-dependent lung tissue, the lung recruitment pressure is calculated with the formula: P = 20 × ΔP / [ΔP - (Pes_insp - Pes_exp)], where the maximum pressure does not exceed 40 cmH₂O. Using the calculated pressure, a single-cycle recruitment maneuver is performed both 30 minutes after pneumoperitoneum establishment and before the end of surgery, each maintained for 10 seconds.
  Other Names: Transpulmonary Pressure; Pleural Pressure
  Arms: Personalized Lung Recruitment Pressure Group
Procedure: Lung Recruitment Maneuver — A single-cycle lung recruitment maneuver was performed at a fixed pressure of 30 cmH₂O for 10 seconds, both 30 minutes after pneumoperitoneum establishmentand immediately before the end of surgery.
  Arms: Fixed Lung Recruitment Pressure Group

SUMMARY:
This is a prospective, single-center, double-blind, randomized controlled trial designed to investigate the individual differences in recruitment efficacy and safety between personalized lung recruitment pressure based on esophageal pressure and conventional fixed lung recruitment pressure. The intervention involved calculating personalized lung recruitment pressure using inspiratory and expiratory esophageal pressures measured via a transnasal esophageal balloon catheter, which was then compared with a fixed pressure of 30 cmH₂O, each applied to maintain a single-cycle lung recruitment maneuver for 10 seconds. A total of 90 patients undergoing elective tracheal intubation under general anesthesia for head-down laparoscopic surgery were randomly assigned to either the experimental or control group. The primary outcome was post-recruitment lung compliance, and secondary outcomes included driving pressure, peak airway pressure (Ppeak), modified LUS score, gas exchange indices, hemodynamic parameters, length of stay in PACU after extubation, incidence of postoperative pulmonary complications (PPCs) on day 3 after surgery, and the rate of non-surgical antibiotic use.

ELIGIBILITY:
Inclusion Criteria:1.Age 18-65 years.2.No restriction on sex.3.ASA physical status classification I-III.4.Scheduled for elective tracheal intubation under general anesthesia in the ead-down (Trendelenburg) position for laparoscopic surgery.5.No recent history of pulmonary infection or respiratory disease, and no prior respiratory-system surgery.

Exclusion Criteria:1.Chronic obstructive pulmonary disease (COPD) or cor pulmonale.2.Poorly controlled chronic diseases such as diabetes mellitus or hypertension.3.Cardiac dysfunction.4.Recent use of non-steroidal anti-inflammatory drugs (NSAIDs) or corticosteroids.5.Esophageal pathology (contraindication to esophageal balloon catheter placement).6.History of esophageal surgery.7.Contraindications to lung recruitment maneuvers: intracranial hypertension, hypovolemic shock, right-heart failure.

-

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2026-02-20 (Estimated); Primary Completion 2026-09-20 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Lung Compliance | From the establishment of pneumoperitoneum until the end of surgery.
  Lung compliance refers to the change in lung volume per unit change in pressure. It was obtained immediately after the lung recruitment maneuver by recording the value displayed on the anesthesia machine.

IPD SHARING:
Plan to Share IPD: No